CLINICAL TRIAL: NCT06406374
Title: Italian Translation and Validation of the Non-Motor Fluctuation Assessment (NoMoFA) Questionnaire.
Brief Title: Italian Translation and Validation of the Non-Motor Fluctuation Assessment (NoMoFA) Questionnaire: an Observational, Multicentric, Cross-sectional, 6-months Duration Study on 200 Consecutive Parkinson's Disease Patients.
Acronym: NoMoFA
Status: Recruiting | Type: Observational
Sponsor: A.O.U. Città della Salute e della Scienza (Other)
Responsible Party: Principal Investigator, Carlo Alberto Artusi, MD, PhD, A.O.U. Città della Salute e della Scienza
Other Study IDs: 0068862
Record Dates: First submitted 2024-05-06; First posted 2024-05-09 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2024-05

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's disease; Non-motor fluctuations; NoMoFA
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Parkinson's disease patients: Patients will present the following inclusion criteria:
  * Diagnosis of idiopathic Parkinson's disease according to the 2015 Movement Disorders Society (MDS) criteria (Postuma et al. Mov Dis, 2015);
  * Italian speaker;
  * Mini-mental state examinations (MMSE) score >25;
  * Presence of symptoms fluctuations, as per a Wearing-off questionnaire 19 (WOQ-19) score>=2;
  * Stable antiparkinsonian medications for at least three months;
  * Ability to provide informed consent.

SUMMARY:
Parkinson's disease (PD) has been traditionally considered a movement disorder. In fact, it is now recognized as a multisystemic disease involving not only the central nervous system and presenting with a constellation of motor and non-motor features. While the dopaminergic therapy used to control motor symptoms can lead to the development of motor fluctuations, characterized by wearing-off, ON-OFF phenomenon, delayed-ON, dose failure, and dyskinesias, it has been demonstrated that also many non-motor symptoms can have daily fluctuations, according to the response to dopaminergic therapy. Therefore, non-motor symptoms may fluctuate in parallel with motor symptoms and their relationship to plasma dopamine concentration, although the exact mechanism of non-motor fluctuations (NMF) remains speculative. Non-motor features tend to worsen during disease progression and prove to severely impact the quality of life of patients, sometimes more than motor symptoms. The Non-Motor Fluctuation Assessment (NoMoFA) Questionnaire is a patient-derived and self-administered questionnaire, recently developed and validated by the International Parkinson and Movement Disorder Society (MDS), that identifies and quantifies the severity of static and fluctuating non-motor symptoms in people with PD. The NoMoFA scale is constituted of a total of 27 items investigating several non-motor features, such as fatigue (the most reported), sleepiness, and confusion. Considering the self-administered nature of the scale, patients must understand the questions, and it should be available in the patient's native language. However, the NoMoFa has not yet been translated into the Italian language. Considering that NoMoFA is a relevant scale in the assessment of patients with PD, we believe it is important to perform a translation and cross-cultural adaptation of the NoMoFA questionnaire in Italian, following the scales translation protocol from the international movement disorders society (MDS), and to analyze the reliability and construct validity of the translated scale in Italian patients with PD who experience non-motor fluctuations. The aim of the study is to translate and validate the adapted Italian version of NoMoFA questionnaire.

DETAILED DESCRIPTION:
This is a multicenter, cross-sectional study involving 200 consecutive patients with a diagnosis of idiopathic PD.

We will collect demographic data such as age, sex and education, and clinical features encompassing age at onset, disease duration, antiparkinsonian treatment, and levodopa-equivalent daily dose (LEDD). Patients will undergo a clinical examination in which we will record the Hoehn and Yahr scale (H&Y) and Movement Disorders Unified Parkinson's Disease Rating Scale (MDS-UPDRS) part I-II- III (in ON state) and IV, and Montreal Cognitive Assessment (MoCA). The answers to the NoMoFA will be obtained giving the self-administered questionnaire to patients during regular follow-up visits. The NoMoFA Questionnaire has a total of 27 items with a total maximum possible score for the NoMoFA of 81 points (27 x 3). To evaluate the stability of the Italian version of the NoMoFA (test-retest reliability), a group of 60 patients will repeat the scale 14 days after the first evaluation.

We will establish a translation team composed of movement disorders specialists who are native speakers of the designated language and fluent in English. As word-for-word translations can be misleading, cultural difference between English and Italian will be taken into account. After translation, a different independent group with same competencies of the first translating team will perform a back-translation. The back-translated version of the rating scale will be compared to the original English version. The translation and back-translation team members in a revised document will fully resolve unclear concepts or ambiguities between the original and back-translated English editions. Before the validation phase, a so-called 'cognitive pretesting' will be performed by submitting the provisional translated scale to 10 PD patients by 2 evaluators external to the translator team. Then, evaluators' and subjects' responses will be integrated into the revisions and retested until all major problems are resolved. Once the translation and cognitive pretesting stages are completed, the translated scale is field-tested in a sample of native speakers of the language of the translated scale (validation).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of idiopathic Parkinson's disease according to the 2015 Movement Disorders Society (MDS) criteria (Postuma et al. Mov Dis, 2015);
* Italian speaker;
* Mini-mental state examinations (MMSE) score >25;
* Presence of symptoms fluctuations, as per a Wearing-off questionnaire 19 (WOQ-19) score>=2;
* Stable antiparkinsonian medications for at least three months
* Ability to provide informed consent.

Exclusion Criteria:

* Atypical Parkinsonian syndrome
* H&Y>4
* Patients under legal protection

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: We will enroll 200 consecutive patients with a diagnosis of idiopathic Parkinson's disease according to validated clinical criteria and experiencing symptoms fluctuations, as per a Wearing-off questionnaire 19 (WOQ-19) score>=2.
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-04-26 (Actual); Primary Completion 2024-06-10 (Estimated); Study Completion 2024-06-10 (Estimated)

PRIMARY OUTCOMES:
Non-motor fluctuations assessment | The entire project is planned for a duration of 13 months.
  The aim of this study is to validate an Italian version of NoMoFA scale for the evaluation of non-motor symptoms fluctuations.

CONTACTS AND LOCATIONS:
Locations (1):
- Dipartimento di Neuroscienze e Salute Mentale SC Neurologia 2U, Torino, TO, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kleiner G, Fernandez HH, Chou KL, Fasano A, Duque KR, Hengartner D, Law A, Margolius A, Poon YY, Saenz Farret M, Saleh P, Vizcarra JA, Stebbins GT, Espay AJ; PSG NoMoFA Study Group. Non-Motor Fluctuations in Parkinson's Disease: Validation of the Non-Motor Fluctuation Assessment Questionnaire. Mov Disord. 2021 Jun;36(6):1392-1400. doi: 10.1002/mds.28507. Epub 2021 Feb 15. PMID 33590555